CLINICAL TRIAL: NCT01032291
Title: A Phase 2, Open-Label Study To Evaluate The Efficacy And Safety Of Lenalidomide In Combination With Cetuximab In Pretreated Subjects With K-Ras Mutant Metastatic Colorectal Cancer
Brief Title: A Study to Assess the Efficacy and Safety of Lenalidomide in Combination With Cetuximab in Pre-treated Patients With KRAS Mutant Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision not to continue with Phase 2b based on non-safety observations during proof of concept phase.
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-COLO-001; 2009-012665-61 (EudraCT Number)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Revlimid; Lenalidomide; Cetuximab; Erbitux; KRAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lenalidomide plus cetuximab (Experimental): Combination therapy of lenalidomide plus cetuximab
  Interventions: Drug: cetuximab; Drug: lenalidomide
- lenalidomide (Experimental): Single agent therapy of lenalidomide
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: cetuximab — Intravenous infusions of cetuximab (400 mg/m^2 Cycle 1 Day 1, thereafter 250 mg/m^2), administered on days 1, 8, 15 and 22 of each 28 day cycle.
  Other Names: Erbitux
  Arms: lenalidomide plus cetuximab
Drug: lenalidomide — Daily oral lenalidomide 25mg on days 1 to 28 of each 28 day cycle
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine whether lenalidomide in combination with cetuximab is safe and effective in patients with KRAS mutant colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic colorectal adenocarcinoma.
2. Confirmed K-RAS mutant tumor
3. Disease progression on oxaliplatin- AND irinotecan-containing regimens, with at least one of these regimens containing bevacizumab.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.

Exclusion Criteria:

1. Use of chemotherapy, hormonal therapy, immunotherapy or any other cancer or experimental treatment ≤ 28 days prior to the first day of the first cycle.
2. Radiotherapy for up to ≥ 30% of the bone marrow.
3. Surgery ≤ 28 days before day 1 of the first cycle (minimally invasive interventions for diagnostic purposes or disease staging are permitted).
4. Previous treatment with cetuximab, panitumumab, pomalidomide (CC-4047), lenalidomide or thalidomide.
5. Untreated, symptomatic brain metastases (brain imaging not required).
6. Venous thromboembolism ≤ 6 months before day1 of the first cycle.
7. Current congestive heart failure (classes II to IV of the New York Heart Association).
8. Myocardial infarction ≤ 12 months before day1 of the first cycle.
9. Uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, M.D., Ph,D, Principal Investigator — Universitaire Ziekenhuis Gasthuisberg K.U. Leuven, Belgium; Josep Tabernero, M.D., Principal Investigator — Hospital Vall d´Hebrón, Servicio de Oncología, Barcelona. Spain
Locations (17):
- Flinders Medical Centre, Dept. of Oncology, Bedford Park, South Australia, Australia
- Belgium (6):
  - UZ Antwerpen Dept. of Medical Oncology, Antwerp
  - ULB Erasme Service de Gastroenterologie, Brussels
  - Grand hôpital de Charleroi, Oncologie, Charleroi
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitaire Ziekenhuis Gasthuisberg K.U. Leuven Gastroenterologie, Oncologie, Leuven
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
- Klinikum Oldenburg gGmbH Klinik für Innere Medizin II, Oldenburg, Lower Saxony, Germany
- Italy (3):
  - Azienda Osperdaliero Universitaria Riuniti Umberto I-GM Lancisi-G. Salesi di Ancona Clinica di Oncologia Medica, Ancona
  - Azienda Ospedaliera Universitaria San Martino Unità Operativa Oncologia Medica, Genova
  - Azienda Ospedaliera Niguarda Ca' Grande, Oncologia Medica Falck, Milan
- Spain (3):
  - Hospital Vall D'Hebron Servicio de Oncología. Unidad de ensayos clínicos, Barcelona
  - Hospital Universitario Marques de Valdecilla Servicio de Oncología, Santander
  - Hospital Clinico Universitario de Valencia Servicio de Oncologia, Valencia
- Sweden (3):
  - Östra Sjukhuset Kirurgkliniken, Gothenburg
  - Karolinska University Hospital, Solna, Karolinska Institutet Dept of Oncology, Stockholm
  - Akademiska Sjukhuset Onkologkliniken, Uppsala

REFERENCES:
- [Derived] Gandhi AK, Shi T, Li M, Jungnelius U, Romano A, Tabernero J, Siena S, Schafer PH, Chopra R. Immunomodulatory effects in a phase II study of lenalidomide combined with cetuximab in refractory KRAS-mutant metastatic colorectal cancer patients. PLoS One. 2013 Nov 11;8(11):e80437. doi: 10.1371/journal.pone.0080437. eCollection 2013. PMID 24244687
- [Derived] Siena S, Van Cutsem E, Li M, Jungnelius U, Romano A, Beck R, Bencardino K, Elez ME, Prenen H, Sanchis M, Sartore-Bianchi A, Tejpar S, Gandhi A, Shi T, Tabernero J. Phase II open-label study to assess efficacy and safety of lenalidomide in combination with cetuximab in KRAS-mutant metastatic colorectal cancer. PLoS One. 2013 Nov 11;8(11):e62264. doi: 10.1371/journal.pone.0062264. eCollection 2013. PMID 24244261

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2b Proof of Concept was designed to enroll 82 participants, however the study terminated early. Forty-three participants were enrolled, however, one was randomized to receive single agent lenalidomide but never received study drug and was excluded from the ITT and Safety populations.
Groups:
- Lenalidomide + Cetuximab (Safety Lead-in): Combination therapy of lenalidomide plus cetuximab during the Safety Lead-in period. Lenalidomide dose of 25 mg/day in combination with cetuximab (IV injections of 400 mg/m^2 first infusion only, then 250 mg/m^2 subsequently administered on Days 1, 8, 15, and 22 of each 28-day cycle).
- Lenalidomide (Proof of Concept): Single agent therapy of lenalidomide (25 mg/day) during the Proof of Concept period.
- Lenalidomide + Cetuximab (Proof of Concept): Combination therapy of lenalidomide plus cetuximab during the Proof of Concept period. Lenalidomide dose of 25 mg/day in combination with cetuximab (IV injections of 400 mg/m^2 first infusion only, then 250 mg/m^2 subsequently administered on Days 1, 8, 15, and 22 of each 28-day cycle).
Period: Safety Lead-in
Arm/Group | Lenalidomide + Cetuximab (Safety Lead-in) | Lenalidomide (Proof of Concept) | Lenalidomide + Cetuximab (Proof of Concept)
Started | 8 | 0 | 0
Completed | 6 (Participants with disease progression) | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: Proof of Concept
Arm/Group | Lenalidomide + Cetuximab (Safety Lead-in) | Lenalidomide (Proof of Concept) | Lenalidomide + Cetuximab (Proof of Concept)
Started | 0 | 22 | 21
Intent to Treat and Safety Populations | 0 | 21 (Participants who took at least one dose of study drug) | 21 (Participants who took at least one dose of study drug)
Completed | 0 | 14 (Participants with disease progression) | 18 (Participants with disease progression)
Not Completed | 0 | 8 | 3
Not completed — Adverse Event | 0 | 5 | 1
Not completed — Death | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Never Received Study Drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide Plus Cetuximab (Safety Lead-In): Combination therapy of lenalidomide plus cetuximab during the Safety Lead-in period. Lenalidomide dose of 25 mg/day in combination with cetuximab (IV injections of 400 mg/m^2 first infusion only, then 250 mg/m^2 subsequently administered on Days 1, 8, 15, and 22 of each 28-day cycle).
- Lenalidomide Plus Cetuximab (Proof of Concept): Combination therapy of lenalidomide plus cetuximab during the Proof of Concept period. Lenalidomide dose of 25 mg/day in combination with cetuximab (IV injections of 400 mg/m^2 first infusion only, then 250 mg/m^2 subsequently administered on Days 1, 8, 15, and 22 of each 28-day cycle).
- Total: Total of all reporting groups
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept) | Total
Number analyzed (Participants) | 8 | 21 | 21 | 50
Age, Customized [Number; unit: participants] — All baseline measures are reported from the safety population.
  participants
    <= 65 years | 7 | 16 | 18 | 41
    >65 years | 1 | 5 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 9 | 22
  Male | 4 | 12 | 12 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White) | 8 | 21 | 20 | 49
  Other (Not Specified) | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Non-Hispanic or Latino | 8 | 21 | 21 | 50
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — The ECOG scale is as follows:
  Grade 0: Fully active, able to carry on all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair.
  participants
    0 | 6 | 10 | 14 | 30
    1 | 2 | 10 | 7 | 19
    2 | 0 | 1 | 0 | 1
    3-5 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicities (DLTs) During the First Treatment Cycle of the Safety Lead-In Period
Description: The number of participants with DLTs determines the maximum tolerated dose of the combination therapy used in the Proof of Concept (POC) period:
  If <2 of the initial 6 participants experience a DLT, then the POC will start with lenalidomide at 25 mg.
  If ≥2 of the initial 6 participants experienced a DLT, then 6 more subjects were to be enrolled at 20 mg lenalidomide.
  If <2 of the additional 6 subjects experienced a DLT, then the lenalidomide starting dose for the POC was to be 20 mg.
  If ≥2 of the additional 6 subjects experienced a DLT, then 6 more subjects were to be enrolled at 15 mg lenalidomide.
  If <2 of the additional 6 subjects experienced a DLT, then the POC was to start with lenalidomide at 15 mg.
  If ≥2 of the additional 6 subjects experienced a DLT, the dosing for the study was to be reassessed by Celgene Corporation and the investigators.
Time Frame: Up to Day 28 (Cycle 1)
Population: All participants who took at least one dose of study medication. If a participant discontinued the study prior to completing the entire first cycle for reasons other than a DLT or if ≥7 days of lenalidomide and/or ≥1 dose of cetuximab were missed during the first cycle for reasons other than a DLT, a replacement would be added at that dose level.
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-in)
Number analyzed (Participants) | 8
participants | 1

2. Post Hoc Outcome: Best Overall Response Assessed by an Independent Review Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1) During the Proof of Concept Period Prior to Early Study Termination
Description: Tumor response was evaluated every 2 cycles beginning with Cycle 3 Day 1 and at treatment discontinuation. Response and progression were evaluated using the RECIST 1.1 criteria (Eisenhauer, 2009).
  * Complete response-disappearance of all lesions
  * Partial response-30% decrease in the sum of diameters of target lesions from baseline
  * Stable disease-neither shrinkage nor increase of lesions.
  * Progressive Disease-20% increase in the sum of diameters of target lesions from nadir.
  Participants with evidence of objective tumor response have the response confirmed with repeat assessments performed at the next scheduled scan.
Time Frame: Week 9 up to week 24
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 21 | 21
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 3 | 5
  Progressive Disease | 13 | 13
  Response Not Evaluable | 5 | 3

3. Secondary Outcome: Kaplan-Meier Estimates for Progression Free Survival (PFS)
Description: PFS was calculated as the time from randomization to the earlier of the first documentation of progressive disease (PD), or death on study due to any cause.
  Analysis was not performed due to the early termination of the study.
Time Frame: up to week 24
Population: Participants who took at least one dose of study treatment. Analysis was not performed due to the early termination of the study.
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Kaplan-Meier Estimates for Duration of Response
Description: Duration of response was defined as the time from the initial response date to progressive disease (PD) for participants who achieved an objective confirmed complete response (CR) or partial response (PR).
  Analysis was not performed due to the early termination of the study.
Time Frame: up to week 24
Population: as for outcome 3
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Disease Control
Description: Known as the Disease Control Rate (DCR), participants with a complete response, partial response or stable disease contribute to the DCR.
  This analysis was not performed due to the early termination of the study.
Time Frame: up to week 24
Population: as for outcome 3
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival
Description: Overall survival was defined as the time between randomization and death. It was intended that participants would be followed for up to 5 years following discontinuation from treatment.
  Analysis was not performed due to the early termination of the study.
Time Frame: up to 5.5 years
Population: as for outcome 3
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: TEAEs are any adverse event occurring or worsening on or after the first treatment of any study drug and within 28 days after the last dose of the last study drug received. Relation to study drug was determined by the investigator. Severity of AE is graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.0. Severity is a 5-point scale: 3= severe or medically significant but not life-threatening 4=life-threatening, urgent intervention required 5=death related to AE.
Time Frame: up to week 28
Population: Participants who took at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Cetuximab (Safety Lead-In) | Lenalidomide (Proof of Concept) | Lenalidomide Plus Cetuximab (Proof of Concept)
Number analyzed (Participants) | 8 | 21 | 21
participants
  >=1 TEAE | 8 | 20 | 21
  Serious TEAE | 5 | 9 | 9
  TEAE leading to discontinuing lenalidomide | 3 | 7 | 5
  TEAE leading to discontinuing cetuximab | 3 | NA — Cetuximab not taken by this treatment arm | 6
  TEAE leading to reduction/interruption of lenalido | 2 | 6 | 9
  TEAE leading to reduction/interruption of cetuxima | 1 | NA — Cetuximab not taken by this treatment arm | 7
  TEAE related to lenalidomide | 5 | 9 | 13
  TEAE related to cetuximab | 8 | NA — Cetuximab not taken by this treatment arm | 19
  TEAE NCI CTC grade 3 or higher | 4 | 13 | 12
  TEAE NCI CTC grade 3+ related to lenalidomide | 3 | 4 | 4
  TEAE NCI CTC grade 3+ related to cetuximab | 2 | NA — Cetuximab not taken by this treatment arm | 7
  Serious TEAE related to lenalidomide | 2 | 0 | 2
  Serious TEAE related to cetuximab | 2 | NA — Cetuximab not taken by this treatment arm | 2

8. Primary Outcome: Percentage of Participants With a Response to Treatment During the Proof of Concept Period
Description: Tumor response was evaluated every 2 cycles beginning with Cycle 3 Day 1 and at treatment discontinuation. Response and progression were evaluated using the RECIST 1.1 criteria (Eisenhauer, 2009).
  Treatment response includes both complete response and partial response.
  * Complete response-disappearance of all lesions
  * Partial response-30% decrease in the sum of diameters of target lesions from baseline
  Analysis was not performed due to the early termination of the study.
Time Frame: week 9 up to week 24
Population: Efficacy Evaluable Population. Analysis was not performed due to the early termination of the study.
Groups:
- Lenalidomide + Cetuximab (Safety Lead-in and Proof of Concept): Combination therapy of lenalidomide plus cetuximab during both the Safety Lead-in and Proof of Concept periods. Lenalidomide dose of 25 mg/day in combination with cetuximab (IV injections of 400 mg/m^2 first infusion only, then 250 mg/m^2 subsequently administered on Days 1, 8, 15, and 22 of each 28-day cycle).
Arm/Group | Lenalidomide (Proof of Concept) | Lenalidomide + Cetuximab (Safety Lead-in and Proof of Concept)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 28 weeks.
Arm/Group | Lenalidomide (Proof of Concept) | Lenalidomide + Cetuximab (Safety Lead-in and Proof of Concept)
Serious Adverse Events (participants affected / at risk) | 9/21 | 14/29
Other Adverse Events (participants affected / at risk) | 16/21 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Proof of Concept) (N=21) | Lenalidomide + Cetuximab (Safety Lead-in and Proof of Concept) (N=29)
Tachycardia (Cardiac disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 2 | 3
Pyrexia (General disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bone Lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Rectal Obstruction (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Extrinsic Vascular Compression (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Proof of Concept) (N=21) | Lenalidomide + Cetuximab (Safety Lead-in and Proof of Concept) (N=29)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 14
Abdominal pain (Gastrointestinal disorders) | 5 | 9
Nausea (Gastrointestinal disorders) | 4 | 10
Constipation (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 4
Ascites (Gastrointestinal disorders) | 2 | 1
Enteritis (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 6 | 11
Asthenia (General disorders) | 6 | 9
Oedema peripheral (General disorders) | 4 | 5
Pyrexia (General disorders) | 3 | 6
Chills (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 2
Xerosis (General disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 2
Paronychia (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Transaminases increased (Investigations) | 2 | 2
Weight decreased (Investigations) | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 3
Polyneuropathy (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 8
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 6
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Enrollment stopped prematurely due to lack of efficacy and failure to achieve the planned response objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication
* Multicenter publication has priority over subset (single center) publication, for duration of 1 year after study completion
* Individual investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 90 days